CLINICAL TRIAL: NCT04987853
Title: Assessment of the Influence of Clinical, Functional, Immunological, and Genetic Factors on the Severity of the Course of Coronavirus Infection With SARS-CoV-2 and Post Covid Syndrome
Brief Title: Clinical, Functional, Immunological and Genetic Factors on the Severity of the Course of Coronavirus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Research Center for Cardiac Surgery, Kazakhstan (Other)
Collaborators: Nazarbayev University Medical Center (Other)
Responsible Party: Principal Investigator, Makhabbat Bekbossynova, Chairman of the Board, National Research Center for Cardiac Surgery, Kazakhstan
Other Study IDs: version 1.0; BR10965164 (Other Grant/Funding Number: MES RK)
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Corona Virus Infection
Keywords: Post Covid syndrome; pneumonia; cardiology; genetic research; immunology
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. blood
  2. deoxyribonucleic acid (DNA) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute COVID patients: Patients in the acute phase of the course of the disease
  Interventions: Diagnostic Test: Clinical and functional analysis; Diagnostic Test: Neurological analysis; Diagnostic Test: Immunological analysis:; Diagnostic Test: Genetic analysis:
- Long Covid Patients: Patients with chronic symptoms after a previous Covid-19 (4-12 weeks)
  Interventions: Diagnostic Test: Clinical and functional analysis; Diagnostic Test: Neurological analysis; Diagnostic Test: Immunological analysis:; Diagnostic Test: Genetic analysis:
- Postcovid patients: Patients with chronic symptoms after a previous Covid-19 (more than 12 weeks)
  Interventions: Diagnostic Test: Clinical and functional analysis; Diagnostic Test: Neurological analysis; Diagnostic Test: Immunological analysis:; Diagnostic Test: Genetic analysis:

INTERVENTIONS:
Diagnostic Test: Clinical and functional analysis — General blood analysis - Complete blood count on an analyzer with differentiation of 5 classes of cells, the ratio of neutrophils to lymphocytes; Blood chemistry - ALT, AST, total bilirubin, direct, LDH, CRP, alpha-amylase, creatinine, urea, glucose, ferritin, glycosylated hemoglobin, vitamin 25 - OH vitamin D, vitamin B12; Coagulogram - D-dimers, fibrinogen, INR, APTT; Other - NT-pro BNP, Homocysteine, IL 6, Troponin, blood group determination; Linked immunosorbent assay - Determination of IgG and IgM antibodies to SARS-CoV-2 coronavirus (COVID-19) in blood serum, RBD; Functional diagnostics • ECG
  * EchoCG + strain
  * CT scan of the lungs
  * Holter
  * SMAD
  * Kidney ultrasound
  * Ultrasound
  * Doppler ultrasonography of veins and arteries
  * Chalder Scale, EQ Questionnaire
  Other Names: Immunological analysis; Genetic analysis
Diagnostic Test: Neurological analysis — Neurological examination with the isolation of neurological syndromes (motor, cognitive impairments, sleep disorders, asthenic-depressive syndromes, etc.).
  2. Neuropsychological methods - research on the scales of anxiety and depression, MMSE, etc.
  3. Instrumental method - EEG, polysonography, ultrasound of the neck vessels, CT perfusion.
  4. Laboratory research methods:
  1. The study of antibodies to some neurospecific antigens - myelin basic protein (MBP), neurospecific enolase (NSE).
  2. Study of cellular immunity (CD3 +, CD4 +, CD8 +) and general indicators of humoral immunity (IgG, IgA, IgM, circulating immune complexes).
Diagnostic Test: Immunological analysis: — A comprehensive immunological analysis will be carried out to determine the level of the immune response. Calculation of the level of CD4 +, CD8 + and NK cells. The level of antibodies of the IgG and IgM classes to the proteins of the coronavirus S1, RBD and N was determined
  Other Names: Multiplex Immunoassay; Immunophenotyping of T-cell and B-cell subpopulations
Diagnostic Test: Genetic analysis: — Isolation (extraction) of DNA will be performed from whole blood using commercial kits according to the manufacturer's instructions. To analyze a large number of genetic markers, it is planned to carry out genome-wide sequencing followed by analysis of genetic polymorphisms of candidate genes encoding coronavirus receptors and immunological factors.

SUMMARY:
The purpose of the program. To determine the clinical, functional, immunological, and genetic factors affecting the severity of the course of acute coronavirus infection COVID-19 and PostCovid syndrome, in order to develop management tactics for such patients to reduce the risk of complications and disability.

DETAILED DESCRIPTION:
Objectives of the program:

1. To determine the clinical and functional characteristics of patients with varying degrees of the course of the acute phase of COVID-19 and Post Covid syndrome.

   1.1. To study the features of neurological disorders in patients with varying degrees of the course of the acute phase of COVID-19 and Post Covid syndrome.
2. To study the immunological profile of patients with varying degrees of the course of the acute phase of COVID-19 and Post Covid syndrome.
3. To study the genetic profile of patients with varying degrees of the course of the acute phase of COVID-19 and Post Covid syndrome.
4. Identify potential predictors of COVID-19 severity.
5. To determine the markers that allows predicting the development of the Post Covid syndrome.
6. Based on the selected markers, develop a COVID-19 outcome scale to determine the tactics of patient management to prevent the development of Post Covid syndrome.

The study will include patients with a positive PCR test for COVID-19. Patients in the acute phase of the course of the disease are monitored and treated in accordance with the republican COVID-19 treatment protocol. After signing the informed consent, the patient will be included in the study. The collection of the necessary materials for subsequent analyzes (clinical-functional, genetic, immunological) will be carried out in accordance with this protocol. Subsequently, patients are observed within one year from the moment of illness in accordance with the study protocol and with the collection of all necessary materials.

Clinical and functional analysis:

Detection of RNA of the COVID-19 virus using PCR analysis. Conducting complex laboratory studies in accordance with table 1.

General blood analysis Complete blood count on an analyzer with differentiation of 5 classes of cells, the ratio of neutrophils to lymphocytes

Blood chemistry ALT, AST, total bilirubin, direct, LDH, CRP, alpha-amylase, creatinine, urea, glucose, ferritin, glycosylated hemoglobin, vitamin 25 - OH vitamin D, vitamin B12

Coagulogram D-dimers, fibrinogen, INR, APTT

Other NT-pro BNP, Homocysteine, IL 6, Troponin, blood group determination

Linked immunosorbent assay Determination of IgG and IgM antibodies to SARS-CoV-2 coronavirus (COVID-19) in blood serum, RBD

Functional diagnostics • ECG

* EchoCG + strain
* CT scan of the lungs
* Holter
* SMAD
* Kidney ultrasound
* Ultrasound
* Doppler ultrasonography of veins and arteries
* Chalder Scale, EQ Questionnaire Table 1. Clinical and functional analysis

Neurological disorders:

1. Neurological examination with the isolation of neurological syndromes (motor, cognitive impairments, sleep disorders, asthenic-depressive syndromes, etc.).
2. Neuropsychological methods - research on the scales of anxiety and depression, MMSE, etc.
3. Instrumental method - EEG, polysonography, ultrasound of the neck vessels, CT perfusion.
4. Laboratory research methods:

   1. The study of antibodies to some neurospecific antigens - myelin basic protein (MBP), neurospecific enolase (NSE).
   2. Study of cellular immunity (CD3 +, CD4 +, CD8 +) and general indicators of humoral immunity (IgG, IgA, IgM, circulating immune complexes).

Immunological analysis:

A comprehensive immunological analysis will be carried out to determine the level of the immune response. Calculation of the level of CD4 +, CD8 + and NK cells. The level of antibodies of the IgG and IgM classes to the proteins of the coronavirus S1, RBD and N was determined Multiplex Immunoassay. For evaluation of immunological parameters, samples are diluted in 200 μl of phosphate buffer, centrifuged and the supernatant analyzed using the manufacturer's protocol. The MILLIPLEX MAP human cytokine / chemokine magnetic bead panel will be used for the analysis of multiple cytokines and chemokines / immunoglobulins, and the Milliplex® magnetic bead panel (HGAMMAG-301K-06, EMD Millipore Corp., Billerica, MA) will be used for immunoglobulin isotyping. Samples will be analyzed on Bioplex BIO-RAD for the following indicators: sCD40L, EGF, Eotaxin / CCL11, FGF-2, Flt-3 ligand, Fractalkine, G-CSF, GM-CSF, GRO, IFN-α2, IFN-γ, IL -1α, IL-1β, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL-17A, IP-10, MCP-1, MCP-3, MDC (CCL22), MIP-1α, MIP-1β, PDGF- AA, PDGF-AB / BB, RANTES, TGF-α, TNF-α, Immunophenotyping of T-cell and B-cell subpopulations using the flow cytometry method. Subpopulations of B- and T-lymphocytes will be examined by staining peripheral blood mononuclear cells (PBMCs) isolated from whole peripheral blood with monoclonal antibodies conjugated to fluorochromes. PBMCs can be isolated from EDTA-treated whole blood using Ficoll density gradient centrifugation or special erythrocyte lysis buffers. It is preferable to analyze isolated PBMCs directly on the day of blood collection, which gives more reliable results. PBMC viability will be assessed using LIVE / DEAD ™ fixed dead cell kits or 0.4% trypan blue and propidium iodide solution. After lysis of erythrocytes and incubation with monoclonal antibodies, the stained cells are resuspended in a staining medium and examined using a MoFlo Astrios flow cytometer (Beckman Coulter, USA). The resulting data will be analyzed using Summit (Beckman Coulter) and FloJo (Tree Star) software.

Forward and side scatter will be used to distinguish the lymphocyte population in addition to the signal from specific fluorochromes. Distribution CD3-, CD5 +, CD19 + (total number of B-lymphocytes), CD5-, CD19 +, CD27 + (memory B-cells), CD19 + CD27- (naive B-cells), CD19 + CD27 + CD38 + IgD - (Class-Switched Memory B-Cells) CD19 + CD27 + CD38 + IgD + (Unswitched Memory B-Cells) will be analyzed on the general lymphocyte population. The distribution of markers CD3, CD4 and CD8 will be analyzed in the pool of T-lymphocytes. To analyze the differentiation status of T cells, cells are additionally stained with anti-CCR7, anti-CD45RO antibodies. Antibodies will be purchased from Invitrogen ™ unless otherwise noted.

Genetic analysis:

Isolation (extraction) of DNA will be performed from whole blood using commercial kits according to the manufacturer's instructions. To analyze a large number of genetic markers, it is planned to carry out genome-wide sequencing followed by analysis of genetic polymorphisms of candidate genes encoding coronavirus receptors and immunological factors.

Sequencing will be performed using high-throughput next generation sequencing platforms Illumina NovaSeq6000 (Illumina), method validation using traditional capillary sequencing - ABI 3730XL ™ DNA Analyzer (Life Technologies), real-time PCR.

Bioinformatic data analysis.Bioinformatics sequencing data will be analyzed. The software packages for bioinformatic analysis of sequencing data (GATK, bwa, bowtie, bowtie2, VarScan etc) will be used. The sequencing data will be compared with the publicly available data from the world's international databases of genomic research (https://www.covid19hg.org/, ExAC, HGMD (Human Gene Mutation Database), ESP, GeneBank, NCBI, ESP6500, 1000Genomes, SNPDb130, Ensembl, ClinVar, SNPedia, etc.). Differences in the type and frequency of genomic variation among the surveyed groups will be determined.

To classify the detected genetic variants, in silico models will be used (SIFT_score / pred, Polyphen2_HDIVscore / pred, Polyphen2_HVAR_score / pred, LRT_score / pred, MutationTaster_score / pred, MutationAssessor_score / pred, FATHMM_score / pred, Radial / MetaRVM_score pred). The classification of clinically significant genetic variants will be carried out according to the international ACMG / AMG criteria.

Statistical analysis:

Statistical analysis will be carried out using version R 3.6.2. Quantitative data, including clinical, biochemical, molecular genetic parameters, will be checked for normality using the Shapiro-Wilks test and recognized as parametric in distribution. Comparison of mean differences will be performed using one-way ANOVA, and subsequent pairwise comparison will be performed using Tukey's special test. Within-group mean differences will be performed using the paired sample t-test. The graphs will be executed using the ggplot2 R package. Statistical analysis will be performed for the multiplex analysis results using the R psych package and standard t-tests.

Inspection frequency:

Patients are followed up for 12 months from the date of illness. Disease detection corresponds to the baseline (day 0). At the time of diagnosis, materials are taken for clinical, functional and immunological diagnostics. After that, the sampling is carried out every month for the next year from the moment of the disease in accordance with the study protocol (Figure 2). The collection of materials for genetic analysis is carried out once.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients with a history of coronavirus infection COVID-19 confirmed by PCR analysis
* Patients who signed informed consent to participate in the study

Exclusion Criteria:

* Refusal to undergo diagnostic procedures determined by the research protocol.
* Evidence for preexisting interstitial lung disease.
* Participation in another study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with a positive PCR test for COVID-19. Patients in the acute phase of the course of the disease are monitored and treated in accordance with the republican COVID-19 treatment protocol. After signing the informed consent, the patient will be included in the study. The collection of the necessary materials for subsequent analyzes (clinical-functional, genetic, immunological) will be carried out in accordance with this protocol. Subsequently, patients are observed within one year from the moment of illness in accordance with the study protocol and with the collection of all necessary materials.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
bioinformatic data analysis | 24 months
  To analyze a large number of genetic markers, it is planned to carry out genome-wide sequencing followed by analysis of genetic polymorphisms of candidate genes encoding coronavirus receptors and immunological factors
the level of the immune response | 24 months
  Calculation of the level of CD4 +, CD8 + and NK cells. The level of antibodies of the IgG and IgM classes to the proteins of the coronavirus S1, RBD and N was determined

CONTACTS AND LOCATIONS:
Overall Officials: Makhabbat Sansyzbaeva, Principal Investigator — Chairman of the Board of "National Research Cardiac Surgery Centre" JSC
Locations (1):
- National Research Center for Cardiac Surgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: all types of supporting information will be shared with the interested party within the framework of the legislation of the Republic of Kazakhstan
URL: http://heartcenter.kz

REFERENCES:
- [Background] Soy M, Keser G, Atagunduz P, Tabak F, Atagunduz I, Kayhan S. Cytokine storm in COVID-19: pathogenesis and overview of anti-inflammatory agents used in treatment. Clin Rheumatol. 2020 Jul;39(7):2085-2094. doi: 10.1007/s10067-020-05190-5. Epub 2020 May 30. PMID 32474885
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. Addendum: A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Dec;588(7836):E6. doi: 10.1038/s41586-020-2951-z. No abstract available. PMID 33199918
- [Result] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Ragab D, Salah Eldin H, Taeimah M, Khattab R, Salem R. The COVID-19 Cytokine Storm; What We Know So Far. Front Immunol. 2020 Jun 16;11:1446. doi: 10.3389/fimmu.2020.01446. eCollection 2020. PMID 32612617
- [Result] Vabret N, Britton GJ, Gruber C, Hegde S, Kim J, Kuksin M, Levantovsky R, Malle L, Moreira A, Park MD, Pia L, Risson E, Saffern M, Salome B, Esai Selvan M, Spindler MP, Tan J, van der Heide V, Gregory JK, Alexandropoulos K, Bhardwaj N, Brown BD, Greenbaum B, Gumus ZH, Homann D, Horowitz A, Kamphorst AO, Curotto de Lafaille MA, Mehandru S, Merad M, Samstein RM; Sinai Immunology Review Project. Immunology of COVID-19: Current State of the Science. Immunity. 2020 Jun 16;52(6):910-941. doi: 10.1016/j.immuni.2020.05.002. Epub 2020 May 6. PMID 32505227
- [Result] Liu J, Wu P, Gao F, Qi J, Kawana-Tachikawa A, Xie J, Vavricka CJ, Iwamoto A, Li T, Gao GF. Novel immunodominant peptide presentation strategy: a featured HLA-A*2402-restricted cytotoxic T-lymphocyte epitope stabilized by intrachain hydrogen bonds from severe acute respiratory syndrome coronavirus nucleocapsid protein. J Virol. 2010 Nov;84(22):11849-57. doi: 10.1128/JVI.01464-10. Epub 2010 Sep 15. PMID 20844028
- [Result] Henderson LA, Canna SW, Schulert GS, Volpi S, Lee PY, Kernan KF, Caricchio R, Mahmud S, Hazen MM, Halyabar O, Hoyt KJ, Han J, Grom AA, Gattorno M, Ravelli A, De Benedetti F, Behrens EM, Cron RQ, Nigrovic PA. On the Alert for Cytokine Storm: Immunopathology in COVID-19. Arthritis Rheumatol. 2020 Jul;72(7):1059-1063. doi: 10.1002/art.41285. Epub 2020 May 10. PMID 32293098
- [Result] Xie X, Zhong Z, Zhao W, Zheng C, Wang F, Liu J. Chest CT for Typical Coronavirus Disease 2019 (COVID-19) Pneumonia: Relationship to Negative RT-PCR Testing. Radiology. 2020 Aug;296(2):E41-E45. doi: 10.1148/radiol.2020200343. Epub 2020 Feb 12. PMID 32049601
- [Result] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Li X, Geng M, Peng Y, Meng L, Lu S. Molecular immune pathogenesis and diagnosis of COVID-19. J Pharm Anal. 2020 Apr;10(2):102-108. doi: 10.1016/j.jpha.2020.03.001. Epub 2020 Mar 5. PMID 32282863
- [Result] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Result] Halpin S, O'Connor R, Sivan M. Long COVID and chronic COVID syndromes. J Med Virol. 2021 Mar;93(3):1242-1243. doi: 10.1002/jmv.26587. Epub 2020 Oct 30. No abstract available. PMID 33034893
- [Result] Mendelson M, Nel J, Blumberg L, Madhi SA, Dryden M, Stevens W, Venter FWD. Long-COVID: An evolving problem with an extensive impact. S Afr Med J. 2020 Nov 23;111(1):10-12. doi: 10.7196/SAMJ.2020.v111i11.15433. PMID 33403997
- [Result] Vink M, Vink-Niese A. Could Cognitive Behavioural Therapy Be an Effective Treatment for Long COVID and Post COVID-19 Fatigue Syndrome? Lessons from the Qure Study for Q-Fever Fatigue Syndrome. Healthcare (Basel). 2020 Dec 11;8(4):552. doi: 10.3390/healthcare8040552. PMID 33322316
- [Derived] Bekbossynova M, Tauekelova A, Kalila Z, Sailybayeva A, Khamitov S, Oralbekova Z. Anxiety and Depression Among Astana Reinfected Patients at 1-, 3-, and 6-Month Follow-Up in the Post-COVID Center. Can Respir J. 2025 Feb 24;2025:5596465. doi: 10.1155/carj/5596465. eCollection 2025. PMID 40041615
- See also: 3. Coronavirus Update (Live): 106,685,660 Cases and 2,327,308 Deaths from COVID-19 Virus Pandemic - Worldometer — https://www.worldometers.info/coronavirus/
- See also: 19. Overview | COVID-19 rapid guideline: managing the long-term effects of COVID-19 | Guidance | NICE — https://www.nice.org.uk/guidance/ng188
- Available data/document: Study Protocol: BR10965164 — https://is.ncste.kz/login
- Available data/document: Informed Consent Form: BR10965164 — https://is.ncste.kz/login
- Available data/document: Clinical Study Report: BR10965164 — https://is.ncste.kz/login

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04987853/Prot_SAP_000.pdf